CLINICAL TRIAL: NCT03998033
Title: An Open-Label, Dose Escalation, Multi-Center Phase I/II Research Trial to Assess the Safety of ET140202 T Cells and Determine the Recommended Phase II Dose ("RP2D") in Adults With Advanced Hepatocellular Carcinoma ("HCC")
Brief Title: Study of ET140202 T Cells in Adults With Advanced Hepatocellular Carcinoma
Acronym: ET-109
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Reallocation of resources to new HCC study.
Sponsor: Eureka Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ETUS18AFPAR109
Record Dates: First submitted 2019-06-07; First posted 2019-06-25 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer; Liver Neoplasm; Metastatic Liver Cancer
Keywords: Hepatocellular Carcinoma; HCC; Advanced HCC; Late-Stage HCC; Liver Cancer; Liver Neoplasm; Metastatic Liver Cancer; Metastatic HCC; T-cell therapy; Immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ET140202 T cells (Experimental): ET140202 Receptor (+) T Cells
  Interventions: Biological: ET140202 autologous T cell product

INTERVENTIONS:
Biological: ET140202 autologous T cell product — Autologous T cells transduced with lentivirus encoding an ET140202 expression construct

SUMMARY:
This is a open-label, dose escalation, multi-center, Phase I / Phase II study to assess the safety of an autologous T-cell product (ET140202) in adult subjects with advanced Alpha-fetoprotein (AFP) positive/Human Leukocyte Antigen (HLA) A-2 positive Hepatocellular Carcinoma (HCC).

DETAILED DESCRIPTION:
The purpose of this study is to investigate a genetically modified autologous T-cell therapy for advanced hepatocellular carcinoma (HCC). ET140202 T cells are autologous T cells genetically modified to carry a TCR-mimic (TCRm) construct capable of mediating cell killing by targeting tumor specific intracellular antigens and addressing solid tumor therapy challenges.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent obtained prior to study procedures
* Histologically confirmed HCC with serum AFP >200ng/ml at time of screening and following most current line of therapy OR radiographic diagnosis of HCC with serum AFP >400ng/ml at time of screening and following most current line of therapy..
* Metastatic or locally advanced, unresectable HCC
* Must have failed or not tolerated, at least one line of systemic therapy for advanced HCC
* Molecular Human Leukocyte Antigen ("HLA") class I allele typing confirms participant carries at least one HLA-A2 allele
* Life expectancy of at least 4 months
* Karnofsky Performance Scale greater than or equal to 70
* At least 1 measurable lesion on imaging by RECIST
* Child-Pugh A or B7
* Absolute neutrophil count greater than or equal to 1,500/mm^3
* Platelet count greater than or equal to 30,000/mm^3

Exclusion Criteria:

* Clinically significant cardiac disease
* Clinically significant pre-existing illness or active infection
* Clinically significant Central Nervous System (CNS) or neural dysfunction
* Active autoimmune disease requiring therapy
* Active malignancy other than HCC unless expected survival is greater than or equal to three years without any treatment (exception: hormone/androgen-depravation therapy) and without any organ involvement
* History of organ transplant
* Compromised circulation in portal vein, hepatic vein, or vena cava due to obstruction
* Advanced HCC involving greater than one-third of the liver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence rates of adverse events (AEs) after infusion of ET140202 T cells | 28 days
  Safety and tolerability of ET140202 T cells as assessed by committee review of dose limiting toxicities (DLTs) and incidence and severity of adverse events (AEs) after infusion
The recommended phase 2 dose (RP2D) regimen of ET140202 T-cell therapy | up to 2 years
  The RP2D will be determined by the study Dose Escalation Committee (DEC) and primarily based on DLT, and secondarily on the best tumor response

SECONDARY OUTCOMES:
Assess efficacy of ET140202 T cells by overall response rate (ORR) using Response Evaluation Criteria In Solid Tumors (RECIST). | up to 2 years
  As a measure of activity, overall response rate will be assessed by radiographic scans and assessed according to RECIST criteria.
Assess efficacy of ET140202 T cells by complete response (CR) using Response Evaluation Criteria In Solid Tumors (RECIST). | up to 2 years
  As a measure of activity, CR rate will be assessed by radiographic scans and assessed according to RECIST criteria.
Assess efficacy of ET140202 T cells by partial response (PR) using Response Evaluation Criteria In Solid Tumors (RECIST). | up to 2 years
  As a measure of activity, PR rate will be assessed by radiographic scans and assessed according to RECIST criteria.
Assess efficacy of ET140202 T cells by progression-free survival (PFS) using Response Evaluation Criteria In Solid Tumors (RECIST). | up to 2 years
  As a measure of activity, PFS rate will be assessed by radiographic scans and assessed according to RECIST criteria.
Assess efficacy of ET140202 T cells by overall survival (OS) using Response Evaluation Criteria In Solid Tumors (RECIST). | up to 2 years
  As a measure of activity, OS rate will be assessed by radiographic scans and assessed according to RECIST criteria.
Assess the expansion of ET140202 T cells in the blood shortly after infusion. | up to 2 years
  The maximum (peak) expansion of ET140202 T cells in the blood post infusion will be determined.
Assess the persistence of ET140202 T cells circulating in blood over time. | up to 2 years
  The level of ET140202 T cells in blood will be determined to assess the persistence of ET140202 T cells during the treatment and follow-up phases of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Eureka Study Director, Study Director — Eureka Therapeutics
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - UC Irvine, Irvine, California
  - UC Davis, Sacramento, California

IPD SHARING:
Plan to Share IPD: No